CLINICAL TRIAL: NCT02283177
Title: A Safety and Tolerability Trial of Crenolanib and Chemotherapy With Cytarabine and Anthracyclines in Patients With Newly Diagnosed Acute Myeloid Leukemia With FLT3 Activating Mutations
Brief Title: A Safety and Tolerability Study of Crenolanib in Combination With Chemotherapy in Newly Diagnosed Acute Myeloid Leukemia Patients With FLT3 Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-006
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Newly Diagnosed AML With FLT3 Activating Mutations
MeSH Terms: interventions — crenolanib; Cytarabine; Daunorubicin; Idarubicin

ARMS (2):
- Cohort A (Experimental): Patients will be given cytarabine and daunorubicin during induction therapy plus crenolanib at 100 mg TID.
  Interventions: Drug: crenolanib; Drug: cytarabine; Drug: daunorubicin
- Cohort B (Experimental): Patients will be given cytarabine and idarubicin during induction therapy plus crenolanib at 100 mg TID.
  Interventions: Drug: crenolanib; Drug: cytarabine; Drug: idarubicin

INTERVENTIONS:
Drug: crenolanib
  Other Names: CP-868,596-26
Drug: cytarabine
Drug: daunorubicin
  Arms: Cohort A
Drug: idarubicin
  Arms: Cohort B

SUMMARY:
This pilot study is designed to evaluate the safety and tolerability of oral crenolanib besylate given sequentially during standard induction and consolidation chemotherapy in patients with newly diagnosed AML with FLT3 activating mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Unequivocal diagnosis of AML based on the WHO classification, excluding acute promyelocytic leukemia
2. No prior therapy for AML, except for hydroxyurea, in this setting is allowed.
3. Subjects with AML evolving from MDS may have received prior MDS therapy with demethylating agents
4. Subjects must have tested positive for FLT3-ITD and/or other FLT3 activating mutations
5. Age ≥18 years
6. ECOG PS 0 - 2
7. Adequate liver function, defined as normal total bilirubin, ALT ≤2.0x ULN, and AST ≤2.0x ULN measured within 24 hours prior to crenolanib commencement
8. Adequate renal function, defined as serum creatinine ≤1.5x ULN or GFR >50 mL/min
9. Negative pregnancy test (serum or urine) for women of childbearing potential (WOCBP)

   • Women considered not of childbearing potential include any of the following: no menses for at least 2 years or menses within 2 years but amenorrheic for at least 2 months and luteinizing hormone (LH) and follicular stimulating hormone (FSH) values within normal range (according to definition of postmenopausal for laboratory used) or bilateral oophorectomy or radiation castration and amenorrheic for at least 3 months or with bilateral tubal ligation
10. WOCBP must practice contraception. Acceptable methods of contraception are double barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, tubal ligations, and abstention
11. Male patients (except those with prior surgical contraceptive procedures) with female partners who are of childbearing potential: Recommendation is for male and partner to use effective contraceptive methods, such as latex condoms, during the study
12. Able and willing to provide written informed consent

Exclusion Criteria:

1. Pre-existing liver diseases (i.e., cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, and sclerosing cholangitis, etc.)
2. Active CNS leukemia
3. Subject with concurrent severe and/or uncontrolled medical conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
4. NYHA Class III-IV heart failure, myocardial infarction <6 months prior to study entry, and/or serious arrhythmia requiring anti-arrhythmic therapy
5. Unable to swallow pills
6. Major surgical procedures within 14 days of administration of crenolanib (does not include line placement as needed for chemotherapy administration).
7. Unwillingness or inability to comply with protocol.
8. Concurrent use of other investigational agents.
9. Subjects who are not eligible for standard chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - City of Hope Medical Center, Duarte, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Wang ES, Goldberg AD, Tallman M, Walter RB, Karanes C, Sandhu K, Vigil CE, Collins R, Jain V, Stone RM. Crenolanib and Intensive Chemotherapy in Adults With Newly Diagnosed FLT3-Mutated AML. J Clin Oncol. 2024 May 20;42(15):1776-1787. doi: 10.1200/JCO.23.01061. Epub 2024 Feb 7. PMID 38324741

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Less Than or Equal to 60 Years of Age: Participants ≤60yrs old who had AML with FLT3 activating mutations received 7+3 induction therapy with cytarabine and either daunorubicin or idarubicin followed by 100 mg crenolanib besylate administered orally three times a day. The participants then received up to four cycles of consolidation chemotherapy with high dose cytarabine followed by 100 mg crenolanib besylate three times a day. Participants not undergoing hematopoietic stem cell transplant received crenolanib for an additional 12 cycles and participants undergoing transplant received 12 cycles of crenolanib post-transplant.
- Participants Greater Than 60 Years of Age: Participants >60yrs old who had AML with FLT3 activating mutations received 7+3 induction therapy with cytarabine and either daunorubicin or idarubicin followed by 100 mg crenolanib besylate administered orally three times a day. The participants then received up to four cycles of consolidation chemotherapy with high dose cytarabine followed by 100 mg crenolanib besylate three times a day. Participants not undergoing hematopoietic stem cell transplant received crenolanib for an additional 12 cycles and participants undergoing transpolant received 12 cycles of crenolanib post-transplant.
Period: Overall Study
Arm/Group | Participants Less Than or Equal to 60 Years of Age | Participants Greater Than 60 Years of Age
Started | 29 | 15
Completed | 28 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants Greater Than 60 Years of Age: Participants >60yrs old who had AML with FLT3 activating mutations received 7+3 induction therapy with cytarabine and either daunorubicin or idarubicin followed by 100 mg crenolanib besylate administered orally three times a day. The participants then received up to four cycles of consolidation chemotherapy with high dose cytarabine followed by 100 mg crenolanib besylate three times a day. Participants not undergoing hematopoietic stem cell transplant received crenolanib for an additional 12 cycles and participants undergoing transplant received 12 cycles of crenolanib post-transplant.
- Total: Total of all reporting groups
Arm/Group | Participants Less Than or Equal to 60 Years of Age | Participants Greater Than 60 Years of Age | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Continuous [Median (Full Range); unit: years] | 51 [19 to 60] | 68 [61 to 75] | 57 [19 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 14 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 15 | 42
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 12 | 34
  Asian | 3 | 2 | 5
  Black or African American | 1 | 1 | 2
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 2 | 0 | 2
FLT3 Mutations [Count of Participants; unit: Participants] — Mutations in the gene encoding the trans-membrane tyrosine kinase FLT3. The type of FLT3 mutation detected by bone marrow assessment at diagnosis was collected. Subjects had either internal tandem duplications (ITD) in the juxtamembrane domain, point mutations or deletions in the tyrosine kinase domain (TKD) or both ITD and TKD mutations together.
  Participants
    ITD only | 23 | 10 | 33
    TKD only | 4 | 4 | 8
    ITD and TKD | 2 | 1 | 3
Cytogenetics [Count of Participants; unit: Participants] — Cytogenetics is the study of the structure and properties of chromosomes. Cytogenetics data was provided by local labs through karyotyping and fluorescent in situ hybridization (FISH). Participants either had normal cytogenetics, abnormal cytogenetics that did not fulfil the definition of complex and abnormal complex cytogenetics. Abnormal cytogenetics represents an irregularity in the number or structure of chromosomes. Complex cytogenetics is defined as the presences of more than or equal to 3 independent abnormalities. Cytogenetics data was not available for 1 participant.
  Participants
    Normal | 21 | 9 | 30
    Abnormal, not complex | 6 | 5 | 11
    Complex | 2 | 0 | 2
    Not Available | 0 | 1 | 1
AML with Antecedent Hematological Disorders [Count of Participants; unit: Participants] — Whether or not subjects had a prior history of antecedent hematological disease. Subjects with de novo AML do not have a history of antecedent hematological disease, while subjects with secondary AML do.
  Participants
    No | 28 | 12 | 40
    Yes | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Crenolanib With Standard Induction Chemotherapy
Description: To determine the response rate to crenolanib. Complete remission (CR) response criteria includes a post-baseline bone marrow (BM) biopsy or aspiration % blasts <5%, the absence of Auer rods and extramedullary leukemia, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L. Complete remission with incomplete blood count recovery (CRi) response includes all CR criteria met, except participant do not achieve either platelet or ANC recovery. Composite Complete CR response includes all subjects who achieve a CR and CRi. Partial Response (PR) response includes all CR criteria met except a decrease of ≥50% in % blasts in the BM aspirate or biopsy from baseline but within 5-25% or bone marrow blasts <5% with persistent Auer rods. Refractory Disease response includes subjects who do not satisfy the criteria for CR, CRi or PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Participants who had AML with FLT3 activating mutations received 7+3 induction therapy with cytarabine and either daunorubicin or idarubicin followed by 100 mg crenolanib besylate administered orally three times a day. The participants then received up to four cycles of consolidation chemotherapy with high dose cytarabine followed by 100 mg crenolanib besylate three times a day. Participants not undergoing hematopoietic stem cell transplant received crenolanib for an additional 12 cycles and participants undergoing transplant received 12 cycles of crenolanib post-transplant.
Arm/Group | Participants Less Than or Equal to 60 Years of Age | Participants Greater Than 60 Years of Age | All Patients
Number analyzed (Participants) | 29 | 15 | 44
Participants
  Composite Complete Remission (CR + CRi) | 26 | 12 | 38
  Complete Remission (CR) | 22 | 12 | 34
  Complete Remission with incomplete count recovery (CRi) | 4 | 0 | 4
  Partial Remission (PR) | 0 | 1 | 1
  Refractory Disease | 3 | 1 | 4
  Not evaluable | 0 | 1 | 1

2. Secondary Outcome: 3-Year Overall Survival
Description: Overall survival (OS) was measured from the date of the first dose of treatment to the date of death from any cause or to the last date that the patient was known to be alive. OS at 3-years is presented.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Less Than or Equal to 60 Years of Age | Participants Greater Than 60 Years of Age | All Patients
Number analyzed (Participants) | 29 | 15 | 44
percentage of participants | 71.4 [56.5 to 90.3] | 33.3 [16.3 to 68.2] | 58 [44.9 to 74.9]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Participants Less Than or Equal to 60 Years of Age | Participants Greater Than 60 Years of Age
All-Cause Mortality (participants affected / at risk) | 9/29 | 10/15
Serious Adverse Events (participants affected / at risk) | 18/29 | 12/15
Other Adverse Events (participants affected / at risk) | 29/29 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Less Than or Equal to 60 Years of Age (N=29) | Participants Greater Than 60 Years of Age (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Cardiac failure (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Bacteraemia (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Less Than or Equal to 60 Years of Age (N=29) | Participants Greater Than 60 Years of Age (N=15)
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 11
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 2
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 3 | 1
Erythema of eyelid (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 3 | 7
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 18 | 12
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Enlarged uvula (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Lip dry (Gastrointestinal disorders) | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 16 | 11
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 3 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 4
Toothache (Gastrointestinal disorders) | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 15 | 7
Asthenia (General disorders) | 0 | 2
Catheter site erythema (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 0 | 1
Catheter site pain (General disorders) | 2 | 2
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 3
Fatigue (General disorders) | 5 | 7
Generalised oedema (General disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 5 | 2
Oedema (General disorders) | 2 | 1
Oedema due to cardiac disease (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 10 | 9
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 8
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Xerosis (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 0
Pneumobilia (Hepatobiliary disorders) | 0 | 1
Graft versus host disease (Immune system disorders) | 1 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0
Graft versus host disease in liver (Immune system disorders) | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 3
Bacterial rhinitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 2 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 3
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Endocarditis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 2 | 0
Hepatic infection fungal (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 3 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 4 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pneumonia fungal (Infections and infestations) | 2 | 3
Pneumonia viral (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Sinusitis fungal (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 6
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood alkaline phosphatase increased (Investigations) | 7 | 5
Blood bilirubin increased (Investigations) | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 4 | 1
Blood testosterone decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Heart rate increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 9
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperlipidaemia (Investigations) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypermagnasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 4
Dysarthria (Nervous system disorders) | 0 | 1
Dysguesia (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 9 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 3
Abnormal dreams (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 7 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 6
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2
Breast mass (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 6
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Embolism venuous (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 1
Hypotension (Vascular disorders) | 3 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 2
Penetrating aortic ulcer (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT02283177/Prot_SAP_000.pdf